CLINICAL TRIAL: NCT01673308
Title: Salvage in Patients With Myelodysplastic Syndrome After Failure of Hypomethylating Agents: Lenalidomide as a Second-line Therapy
Brief Title: Lenalidomide After Failure of Hypomethylating Agents in Myelodysplastic Syndrome
Acronym: VIOLET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ulsan University Hospital (Other)
Collaborators: Cooperative Study Group A for Hematology (Network)
Responsible Party: Principal Investigator, Hawk Kim, Associate Professor, Ulsan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MDS-PI-0722
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Lenalidomide treatment arm
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 10 mg orally on days 1 to 21 of a 28-day cycle for at least 4 cycles until intolerance or disease progression.
  Other Names: Revlimid

SUMMARY:
This is a Phase II study to evaluate the efficacy of second-line lenalidomide monotherapy for myelodysplastic syndrome (MDS) patients who failed to hypomethylating agents.

DETAILED DESCRIPTION:
There is no standard therapy after the failure of hypomethylating agents only providing supportive cares including transfusion or cytokine therapies. Lenalidomide is the treatment of choice in case of MDS with 5q deletion. A study of lenalidomide for non-5q deletion MDS patients showed that transfusion independency rate was 26% which was relatively acceptable and suggested that lenalidomide could be used for non-5q deletion MDS patients. There is no datum for second-line lenalidomide therapy after hypomethylating agents. MDS which has highly complex pathogenesis backgrounds will have distinctive subtype for each therapy and each treatment drug can have distinctive subgroup for the response. In fact the investigators don't know which patient will be responsive hypomethylating agents or lenalidomide except for 5q deletion. This suggests that second line therapy after the first line failure in MDS will be different with other type of relapsed/refractory disease which will be tend to more resistant to subsequent therapies. In this regard, there is a possibility to have a relatively high response rate to second line lenalidomide in this selected subset who has failed to the hypomethylation therapy or some patients will be responsive regardless of treatment line. Recent data suggested that MDS with JAK2 mutation will be responsive to lenalidomide. The investigators will analyze the JAK2 mutation status in response evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome by world health organization (WHO) classification
* Treatment failure after hypomethylating agents (HMA; azacitidine or decitabine); Intolerant to hypomethylating agents or Progressive disease after HMA
* Age over 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate organ function (serum creatinine ≤ 2.5 mg/dL, serum aspartate transaminase or alanine transaminase ≤ 3.0 x upper limit of normal (ULN), and serum direct bilirubin ≤ 2.0 mg/dL).

Exclusion Criteria:

* Previous therapy history for MDS except for hypomethylating agents, cytokines (granulocyte-stimulating agents or erythropoietin) or supportive care.
* Patients who cannot keep the strict contraception or who willing to be pregnant.
* Contraindication to lenalidomide: Females who are or may become pregnant; Lenalidomide is contraindicated in any patients who have demonstrated hypersensitivity to the drug or its components; Lenalidomide capsules contain lactose. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take this medicinal product.
* Patients who cannot take lenalidomide orally
* Current enrollment to other clinical trial
* Presence of uncontrolled bleeding
* Severe or life-threatening other medical conditions
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* History of congenital or acquired coagulopathy unrelated to malignancy
* History of non-compliance or patient who cannot sign informed consent
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)
* Candidate of hematopoietic stem cell transplantation who cannot complete 4 cycles of lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Response criteria by international working group (IWG) 2006 criteria | 12 months

SECONDARY OUTCOMES:
Safety | 2 years
  Safety assessed by national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, M.D., Ph.D., Principal Investigator — Ulsan University Hospital, University of Ulsan College of Medicine
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

REFERENCES:
- [Background] Prebet T, Gore SD, Esterni B, Gardin C, Itzykson R, Thepot S, Dreyfus F, Rauzy OB, Recher C, Ades L, Quesnel B, Beach CL, Fenaux P, Vey N. Outcome of high-risk myelodysplastic syndrome after azacitidine treatment failure. J Clin Oncol. 2011 Aug 20;29(24):3322-7. doi: 10.1200/JCO.2011.35.8135. Epub 2011 Jul 25. PMID 21788559
- [Background] Jabbour E, Garcia-Manero G, Batty N, Shan J, O'Brien S, Cortes J, Ravandi F, Issa JP, Kantarjian H. Outcome of patients with myelodysplastic syndrome after failure of decitabine therapy. Cancer. 2010 Aug 15;116(16):3830-4. doi: 10.1002/cncr.25247. PMID 20564137
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420
- [Background] Ades L, Boehrer S, Prebet T, Beyne-Rauzy O, Legros L, Ravoet C, Dreyfus F, Stamatoullas A, Chaury MP, Delaunay J, Laurent G, Vey N, Burcheri S, Mbida RM, Hoarau N, Gardin C, Fenaux P. Efficacy and safety of lenalidomide in intermediate-2 or high-risk myelodysplastic syndromes with 5q deletion: results of a phase 2 study. Blood. 2009 Apr 23;113(17):3947-52. doi: 10.1182/blood-2008-08-175778. Epub 2008 Nov 5. PMID 18987358
- [Background] Jadersten M, Hellstrom-Lindberg E. Myelodysplastic syndromes: biology and treatment. J Intern Med. 2009 Mar;265(3):307-28. doi: 10.1111/j.1365-2796.2008.02052.x. Epub 2008 Dec 17. PMID 19141095
- [Background] Heise C, Carter T, Schafer P, Chopra R. Pleiotropic mechanisms of action of lenalidomide efficacy in del(5q) myelodysplastic syndromes. Expert Rev Anticancer Ther. 2010 Oct;10(10):1663-72. doi: 10.1586/era.10.135. PMID 20942636
- [Background] Nomdedeu M, Maffioli M, Calvo X, Martinez-Trillos A, Baumann T, Diaz-Beya M, Aguilar JL, Rozman M, Costa D, Esteve J, Cervantes F, Colomer D, Nomdedeu B. Efficacy of lenalidomide in a patient with myelodysplastic syndrome with isolated del(5q) and JAK2V617F mutation. Leuk Res. 2011 Sep;35(9):1276-8. doi: 10.1016/j.leukres.2011.06.008. Epub 2011 Jul 20. No abstract available. PMID 21764129
- [Background] Raza A, Reeves JA, Feldman EJ, Dewald GW, Bennett JM, Deeg HJ, Dreisbach L, Schiffer CA, Stone RM, Greenberg PL, Curtin PT, Klimek VM, Shammo JM, Thomas D, Knight RD, Schmidt M, Wride K, Zeldis JB, List AF. Phase 2 study of lenalidomide in transfusion-dependent, low-risk, and intermediate-1 risk myelodysplastic syndromes with karyotypes other than deletion 5q. Blood. 2008 Jan 1;111(1):86-93. doi: 10.1182/blood-2007-01-068833. Epub 2007 Sep 24. PMID 17893227
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072